CLINICAL TRIAL: NCT01161524
Title: A Randomized, Double-blind, Placebo-controlled, Parallel-group Study With an Open-label Extension Phase to Evaluate the Effect of Perampanel (E2007) on Cognition, Growth, Safety, Tolerability, and Pharmacokinetics When Administered as an Adjunctive Therapy in Adolescents (12 to Less Than 18 Years of Age) With Inadequately Controlled Partial-onset Seizures
Brief Title: A Study With an Open-label Extension Phase to Evaluate the Effect of Perampanel (E2007) on Cognition, Growth, Safety, Tolerability, and Pharmacokinetics in Adolescents
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eisai Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: E2007-G000-235
Record Dates: First submitted 2010-07-12; First posted 2010-07-13 (Estimated); Results first posted 2019-05-15 (Actual); Last update posted 2019-05-15 (Actual); Status verified 2015-11

CONDITIONS: Epilepsy
MeSH Terms: conditions — Epilepsy | interventions — perampanel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Perampenal (Core Study) (Experimental): Participants received perampanel 2 mg per day and up-titrated weekly in 2-mg increments to a target dose range of 8 to 12 mg per day.
  Interventions: Drug: Perampanel
- Placebo (Core Study) (Placebo Comparator): Participants received matching placebo tablets once a day (6 tablets of placebo).
  Interventions: Drug: Placebo
- Perampanel (Extension Phase) (Experimental): During the Extension Phase, participants previously assigned to perampanel arm (Core Study) continued taking study medication at the dose achieved at the end of the Core Study once daily. Participants previously assigned to a placebo arm (Core Study) started perampanel dose at 2 mg/day and up-titrated weekly in 2-mg increments up to a maximum dose of 12 mg/day.
  Interventions: Drug: Perampanel

INTERVENTIONS:
Drug: Perampanel — 2 mg titrated up to 8-12 mg maximum; taken once daily.
  Arms: Perampanel (Extension Phase); Perampenal (Core Study)
Drug: Placebo — Matching Placebo taken once daily.
  Arms: Placebo (Core Study)

SUMMARY:
This study is designed to investigate the short- and long-term effects of perampanel on cognition, growth, and development in adolescents.

DETAILED DESCRIPTION:
This study consisted of the Core Study and the Extension Part A and B. The Core Study consisted of 2 phases: Prerandomization and Randomization. The Prerandomization Phase lasted up to 1 week, during which participants were assessed for their eligibility to participate in the study. The Randomization Phase consisted of 3 periods: Titration (6 weeks), Maintenance (13 weeks), and Follow-up (4 weeks; only for those participants not rolling over into the Extension Phase). During the Core Study Titration and Maintenance Periods, participants were randomized into perampanel (2 to 12 mg per day) or placebo treatment groups in a 2:1 ratio within each of the age-matched categories (ie, greater than or equal to 12 to less than 15 and greater than or equal to 15 to less than 18).

The extension phase consisted of part A (Conversion Period - 6 weeks and Maintenance period - 25 weeks) and Part B (Optional Extension Phase -52 weeks). The maximum duration for participation in Part B was 52 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Considered reliable and willing to be available for the study duration and was able to record seizures and report adverse events (AEs) themselves or had a legal guardian or a caregiver who could record seizures and report AEs for them.
2. Understand the requirements of the Cognitive Drug Research (CDR) System tests and able to perform the tests appropriately at Visit 1.
3. Male or female, 12 to less than 18 years of age at the time of consent/assent
4. Had a diagnosis of epilepsy with partial-onset seizures with or without secondarily generalized seizures according to the International League Against Epilepsy's (ILAE) Classification of Epileptic Seizures (1981).
5. Diagnosis was established at least 6 months prior to Visit 1, by clinical history and an electroencephalogram (EEG) that was consistent with localization-related epilepsy; normal interictal EEGs were allowed provided that the subject met the other diagnosis criterion (ie, clinical history).
6. Had a brain imaging (e.g., magnetic resonance imaging [MRI] scan or computed tomography [CT]) within the 5 years prior to Visit 1 that ruled out a progressive cause of epilepsy.
7. Had at least 1 partial-onset seizure during the 4 weeks prior to Visit 1 despite a stable regimen of 1 to 3 concomitant antiepileptic drugs (AEDs).
8. Were currently being treated with stable doses of 1-3 AEDs. Only 1 inducer AED (either carbamazepine or phenytoin) out of the maximum of 3 AEDs was allowed.
9. Were on a stable dose of the same concomitant AED(s) for at least 4 weeks prior to Visit 1; in the case where a new AED regimen was initiated for a subject, the dose must have been stable for at least 8 weeks prior to Visit 1.
10. Female subjects of childbearing potential must had a negative serum human chorionic gonadotropin (beta-hCG) at Visit 1 and a negative urine pregnancy test prior to randomization at Visit 2. Female subjects of period of at least 60 days following administration of the last dose of study medication to commit to the consistent and correct use of a medically acceptable method of birth control (e.g., a double-barrier method [condom + spermicide, condom + diaphragm with spermicide]). Abstinence was considered an acceptable method of contraception on a case by case basis upon prior approval by the Medical Monitor.
11. Had an intelligence quotient (IQ) of greater than or equal to 70, using the Kaufman Brief Intelligence Test, second edition (KBIT-2).
12. Provided written informed consent signed by the legal guardian and a written assent from the subject prior to entering the study or undergoing any study procedures.

Extension Phase:

Had completed all scheduled visits up to and including Visit 8 in the Core Study Randomization Phase.

Exclusion Criteria:

1. Had a diagnosis of primary generalized epilepsies or seizures such as absences and/or myoclonic epilepsies.
2. Had current or a history of pseudo-seizures (psychogenic non-epileptic seizures [PNES]) within approximately 5 years prior to Visit 1.
3. Had a diagnosis of Lennox-Gastaut syndrome.
4. Had seizure clusters where individual seizures could not be counted.
5. Had a history of status epilepticus that required hospitalization during the 12 months prior to the Visit 1.
6. Had an unstable psychiatric diagnosis that could confound the investigator's ability to conduct the study or that could prevent completion of the protocol specified tests (e.g., significant suicide risk, including suicidal behavior and ideation 6 months prior to Visit 1, current psychotic disorder, or acute mania).
7. Had any concomitant illnesses/co-morbidities (e.g., autism, attention deficit hyperactivity disorder [ADHD]) at Visit 1 that could severely affect cognitive function during the course of the study.
8. Had previously participated in a clinical trial involving perampanel.
9. Had chronically or routinely use benzodiazepines and who have not discontinued the use at least 4 weeks prior to Visit 1.

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 133 (Actual)
Dates: Start 2010-09 (Actual); Primary Completion 2013-06 (Actual); Study Completion 2014-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Haichen Yang, M.D., M.A., Study Director — Study Director
Locations (37):
- United States (11):
  - Aurora, Colorado
  - Gulf Breeze, Florida
  - Orlando, Florida
  - Tampa, Florida
  - Indianapolis, Indiana
  - Chesterfield, Missouri
  - Gibbsboro, New Jersey
  - Akron, Ohio
  - Memphis, Tennessee
  - Nashville, Tennessee
  - Dallas, Texas
- Heidelberg, Victoria, Australia
- Belgium (3):
  - Brussels
  - Leuven
  - Ottignies
- Ostrava, Czechia
- Hungary (3):
  - Budapest
  - Debrecen
  - Miskolc
- India (7):
  - Bangalore
  - Hyderabad
  - Mangalore
  - Nagpur
  - New Delhi
  - Pune
  - Secunderabad
- Latvia (3):
  - Daugavpils
  - Riga
  - Valmiera
- Poland (2):
  - Gdansk
  - Poznan
- South Korea (2):
  - Daegu
  - Seoul
- Spain (2):
  - Madrid, Madrid, Communidad de
  - Valencia, Valencia
- Thailand (2):
  - Bangkok
  - Nonthaburi

REFERENCES:
- [Derived] Bresnahan R, Hill RA, Wang J. Perampanel add-on for drug-resistant focal epilepsy. Cochrane Database Syst Rev. 2023 Apr 14;4(4):CD010961. doi: 10.1002/14651858.CD010961.pub2. PMID 37059702
- [Derived] Pina-Garza JE, Lagae L, Villanueva V, Renfroe JB, Laurenza A, Williams B, Kumar D, Meador KJ. Long-term effects of adjunctive perampanel on cognition in adolescents with partial seizures. Epilepsy Behav. 2018 Jun;83:50-58. doi: 10.1016/j.yebeh.2018.03.029. Epub 2018 Apr 10. PMID 29653338
- [Derived] Meador KJ, Yang H, Pina-Garza JE, Laurenza A, Kumar D, Wesnes KA. Cognitive effects of adjunctive perampanel for partial-onset seizures: A randomized trial. Epilepsia. 2016 Feb;57(2):243-51. doi: 10.1111/epi.13279. Epub 2016 Jan 1. PMID 26724782

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of the 154 participants screened for entry into the Core Study, 21 were screen failures and 133 were randomized and treated. A total of 119 participants completed the Core Study, and 114 participants entered the Extension Phase.
Groups:
- Perampanel (Core Study): Participants received perampanel 2 mg per day and up-titrated weekly in 2-mg increments to a target dose range of 8 to 12 mg per day.
Period: Core Study (23 Weeks)
Arm/Group | Perampanel (Core Study) | Placebo (Core Study) | Perampanel (Extension Phase)
Started | 85 | 48 | 0
Completed | 76 | 43 | 0
Not Completed | 9 | 5 | 0
Not completed — Adverse Event | 3 | 0 | 0
Not completed — Other | 1 | 0 | 0
Not completed — Withdrawal of Consent | 1 | 1 | 0
Not completed — Lost to Follow-up | 1 | 2 | 0
Not completed — Subject Choice | 3 | 2 | 0
Period: Extension Phase (Approximately 83 Weeks)
Arm/Group | Perampanel (Core Study) | Placebo (Core Study) | Perampanel (Extension Phase)
Started | 0 | 0 | 114
Completed | 0 | 0 | 90
Not Completed | 0 | 0 | 24
Not completed — Adverse Event | 0 | 0 | 8
Not completed — Other | 0 | 0 | 6
Not completed — Lost to Follow-up | 0 | 0 | 1
Not completed — Subject Choice | 0 | 0 | 5
Not completed — Inadequate Therapeutic Effect | 0 | 0 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Perampenal (Core Study) | Placebo (Core Study) | Total
Number analyzed (Participants) | 85 | 48 | 133
Age, Continuous [Mean (Standard Deviation); unit: Years] | 14.3 (1.74) | 14.3 (1.88) | 14.3 (1.79)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33 | 20 | 53
  Male | 52 | 28 | 80
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 1 | 3
  Not Hispanic or Latino | 82 | 47 | 129
  Unknown or Not Reported | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to Week 19 in Cognition Drug Research (CDR) System Global Cognition Score (Core Study)
Description: The CDR System Global Cognitive score was derived from the average of 5 CDR System cognitive domain scores (Power of Attention, Continuity of Attention, Quality of Episodic Memory, Quality of Working Memory, and Speed of Memory). The domain scores were normalized to mean of 50 and standard deviation of 10 before taking the average. The scale ranged from 0 - 100. An increase in the Global Cognitive Score indicates improvement, while a decrease indicates worsening in cognitive function.
Time Frame: Baseline (Visit 2/Week 0 Evaluation) and Week 19 LOCF (last observation carried forward)
Population: Full Analysis Set (FAS) for Cognition: All randomized subjects who received study drug, had baseline cognition data, and had at least one postdose CDR System cognitive battery test assessments at or after Week 10.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Perampanel (Core Study) | Placebo (Core Study)
Number analyzed (Participants) | 79 | 44
Scores on a scale | -1.0 (8.86) | 1.1 (7.14)

2. Secondary Outcome: Change From Baseline at Week 19 in the Power of Attention T-score in the Randomization Phase (Core Study)
Description: The Power of Attention domain (one of the 5 CDR System cognitive domains) was a measure of focused attention and information processing, comprised of the 3 CDR System attention tasks: the simple reaction time, choice reaction time and digit vigilance tasks. Z-scores were calculated for each domain by subtracting each participant's domain score from the normative population mean of that domain and dividing the result by the standard deviation (SD) of the normative population mean. Z-scores were converted into T-scores by multiplying by 50 and adding 50. Power of Attention were also multiplied by -1, so that for all domains, greater T-scores reflected superior cognitive function. T-scores ranged from 0 to 100, with a mean of 50 and an SD of 10. The CDR System Global Cognition score was created by adding the T-scores for the five domains. A decrease in the score of Power of Attention indicated improvement in cognitive function and a negative change reflects impairment from baseline.
Time Frame: Baseline and Week 19
Population: FAS for cognition (Core Study)
Measure: Least Squares Mean (Standard Error); unit: T-score
Arm/Group | Perampanel (Core Study) | Placebo (Core Study)
Number analyzed (Participants) | 79 | 44
T-score | -6.9 (2.3) | -2.7 (3.0)

3. Secondary Outcome: Change From Baseline at Week 19 in the Continuity of Attention T-score in the Randomization Phase (Core Study)
Description: The Continuity of Attention domain (one of the 5 CDR System cognitive domains) was a measure of sustained attention, comprised of the accuracy scores from 2 of the CDR System attention tasks: choice reaction time and digit vigilance. Z-scores were calculated for this domain using normative data from the CDR System database for the age range of the study population. Specifically, Z-scores were calculated by subtracting each participant's domain score from the normative population mean of that domain and dividing the result by the SD of the normative population mean. Z-scores were converted into T-scores by multiplying by 50 and adding 50. Greater T-scores reflected superior cognitive function and a negative change from baseline reflects impairment compared to baseline. T-scores ranged from 0 to 100, with a mean of 50 and an SD of 10.
Time Frame: Baseline and Week 19
Population: FAS for cognition (Core Study)
Measure: Least Squares Mean (Standard Error); unit: T-score
Arm/Group | Perampanel (Core Study) | Placebo (Core Study)
Number analyzed (Participants) | 79 | 44
T-score | -1.7 (0.9) | 1.6 (1.2)

4. Secondary Outcome: Change From Baseline at Week 19 in the Quality of Episodic Secondary Memory T-score in the Randomization Phase (Core Study)
Description: The Quality of Episodic Secondary Memory domain was a measure of the capability of individuals to encode, store, and subsequently retrieve verbal and nonverbal information in episodic (or declarative) memory; what was meant by memory in everyday terminology. This measure was derived by summing the scores from the 4 tasks: immediate and delayed word recall, word recognition, and picture recognition. Z-scores were calculated by subtracting each participant's domain score from the normative population mean of that domain and dividing the result by the SD of the normative population mean. Z-scores were converted into T-scores by multiplying by 50 and adding 50. Greater T-scores reflected superior cognitive function. T-scores ranged from 0 to 100, with a mean of 50 and an SD of 10. A high score reflects a good ability to store, hold and retrieve information of an episodic nature (i.e. an event or a name) and a negative change from baseline reflects impairment compared to baseline.
Time Frame: Baseline and Week 19
Population: FAS for cognition (Core Study)
Measure: Least Squares Mean (Standard Error); unit: T-score
Arm/Group | Perampanel (Core Study) | Placebo (Core Study)
Number analyzed (Participants) | 79 | 44
T-score | 3.0 (1.1) | -1.2 (1.5)

5. Secondary Outcome: Change From Baseline at Week 19 in the Quality of Working Memory (Short Term) T-score in the Randomization Phase (Core Study)
Description: The Quality of Working Memory domain (one of the 5 CDR System cognitive domains) was a measure of reflecting how well individuals can hold numeric and spatial information 'on line' in working memory. Z-scores were calculated by subtracting each participant's domain score from the normative population mean of that domain and dividing the result by the SD of the normative population mean. Z-scores were converted into T-scores by multiplying by 50 and adding 50. Greater T-scores reflected superior cognitive function. T-scores ranged from 0 to 100, with a mean of 50 and an SD of 10. A higher score reflects a good working memory and a negative change from baseline reflects impairment compared to the baseline assessment.
Time Frame: Baseline and Week 19
Population: FAS for cognition (Core Study)
Measure: Least Squares Mean (Standard Error); unit: T-score
Arm/Group | Perampanel (Core Study) | Placebo (Core Study)
Number analyzed (Participants) | 79 | 44
T-score | 1.1 (1.2) | 2.0 (1.5)

6. Secondary Outcome: Change From Baseline at Week 19 in the Speed of Memory T-score in the Randomization Phase (Core Study)
Description: The Speed of Memory domain (one of the 5 CDR System cognitive domains) was a measure, which reflects the time taken to accurately retrieve information from working and episodic memory. Z-scores were calculated for this domain using normative data from the CDR System database for the age range of the study population. Specifically, Z-scores were calculated by subtracting each participant's domain score from the normative population mean of that domain and dividing the result by the SD of the normative population mean. Z-scores were converted into T-scores by multiplying by 50 and adding 50. Speed of Memory were also multiplied by -1, so that for all domains, greater T-scores reflected superior cognitive function and a negative change from baseline reflects impairment compared to the baseline assessment. T-scores ranged from 0 to 100, with a mean of 50 and an SD of 10.
Time Frame: Baseline and Week 19
Population: FAS for cognition (Core Study)
Measure: Least Squares Mean (Standard Error); unit: T-score
Arm/Group | Perampanel (Core Study) | Placebo (Core Study)
Number analyzed (Participants) | 79 | 44
T-score | 0.3 (2.1) | 7.0 (2.7)

7. Secondary Outcome: Percentage of Participants Who Experienced 50% or More Decrease in Seizure Frequency (Core Study)
Description: A responder was a participant who experienced a 50% or greater reduction in seizure frequency compared to the baseline of the Randomization Phase.
Time Frame: From Baseline up to Week 19 LOCF
Population: FAS for Efficacy: All subjects who sign informed consent, were randomized, received treatment, and had at least one postdose seizure efficacy assessment in seizure record was included in this analysis set.
Measure: Number; unit: Percentage of Participants
Arm/Group | Perampanel (Core Study) | Placebo (Core Study)
Number analyzed (Participants) | 83 | 46
Percentage of Participants | 53.0 | 34.8

8. Secondary Outcome: Percent Change From Baseline in Seizure Frequency Per 28 Days During the Treatment Duration of the Randomization Phase (Core Study)
Description: Seizure frequency was based on overall number of seizures obtained by summing the 4 seizure types (all partial seizure types, that is, simple partial without motor signs, simple partial with motor signs, complex partial, and complex partial with secondary generalization) collected via the patient diary over a particular time interval and re-scaled to 28 days window.
Time Frame: Baseline and Week 19 LOCF
Population: FAS for efficacy
Measure: Median (Full Range); unit: Percent change
Arm/Group | Perampanel (Core Study) | Placebo (Core Study)
Number analyzed (Participants) | 83 | 46
Percent change | -58.0 [-100.0 to 3404.0] | -24.0 [-100.0 to 644.7]

9. Secondary Outcome: Number of Participants Who Achieved Seizure-Free Status During the Maintenance Period and the Last 28 Days of the Maintenance Period During the Randomization Phase (Core Study)
Description: Number of Participants who were seizure free, were assessed.
Time Frame: 13 Week Maintenance Period
Population: FAS for efficacy
Measure: Number; unit: Participants
Arm/Group | Perampanel (Core Study) | Placebo (Core Study)
Number analyzed (Participants) | 83 | 46
Participants
  Complete Maintenance Period | 18 | 7
  Last 28 Days of Maintenance Period | 31 | 13

10. Secondary Outcome: Percent Change From Baseline in Seizure Frequency Per 28 Days Over the Perampanel Duration Exposure (Extension Phase)
Description: The median percent change in total partial onset seizure frequency per 28 days during the Extension Phase relative to the Pre-perampanel Baseline from Week 1 of perampanel treatment through successive 13-week intervals (Weeks 1 to 13 for subjects with any data, Weeks 1 to 26 for subjects with exposure of more than 13 weeks, Weeks 1 to 39 for subjects with exposure of more than 26 weeks, and Week 1 to 52 for subjects with exposure of more than 52 weeks) are presented. The perampanel exposure duration starts from the first perampanel dose (in the Core Study for subjects previously randomized to perampanel or Extension Phase for subjects previously randomized to placebo) to the last perampanel dose in the Extension Phase.
Time Frame: Week 1-13, Week 14-26, Week 27-39, and Week 40-52
Population: The Full Analysis Set (FAS) for Efficacy: All participants who received study drug during the Extension Phase, had baseline seizure frequency data, and had at least one observation of valid seizure diary data during the Extension Phase.
Measure: Median (Full Range); unit: Percent change
Arm/Group | Perampanel (Extension Phase)
Number analyzed (Participants) | 114
Percent change
  Week 1-13 (any exposure duration); N=114 | -59.1 [-100.0 to 2909.6]
  Week 1-13 (at least 13 weeks of exposure); N=109: number analyzed (Participants) | 109
  Week 1-13 (at least 13 weeks of exposure); N=109 | -60.4 [-100.0 to 2909.6]
  Week 1-13 (at least 26 weeks of exposure); N=107: number analyzed (Participants) | 107
  Week 1-13 (at least 26 weeks of exposure); N=107 | -60.9 [-100.0 to 2909.6]
  Week 1-13 (at least 39 weeks of exposure); N=90: number analyzed (Participants) | 90
  Week 1-13 (at least 39 weeks of exposure); N=90 | -54.2 [-100.0 to 2909.6]
  Week 1-13 (at least 52 weeks of exposure); N=67: number analyzed (Participants) | 67
  Week 1-13 (at least 52 weeks of exposure); N=67 | -60.9 [-100.0 to 2909.6]
  Week 14-26 (at least 26 weeks of exposure); N=107: number analyzed (Participants) | 107
  Week 14-26 (at least 26 weeks of exposure); N=107 | -63.7 [-100.0 to 4108.2]
  Week 14-26 (at least 39 weeks of exposure); N=90: number analyzed (Participants) | 90
  Week 14-26 (at least 39 weeks of exposure); N=90 | -58.8 [-100.0 to 4108.2]
  Week 14-26 (at least 52 weeks of exposure); N=67: number analyzed (Participants) | 67
  Week 14-26 (at least 52 weeks of exposure); N=67 | -61.3 [-100.0 to 4108.2]
  Week 27-39 (at least 39 weeks of exposure); N=90: number analyzed (Participants) | 90
  Week 27-39 (at least 39 weeks of exposure); N=90 | -73.1 [-100.0 to 792.3]
  Week 27-39 (at least 52 weeks of exposure); N=67: number analyzed (Participants) | 67
  Week 27-39 (at least 52 weeks of exposure); N=67 | -74.1 [-100.0 to 792.3]
  Week 40-52 (at least 52 weeks of exposure); N=53: number analyzed (Participants) | 53
  Week 40-52 (at least 52 weeks of exposure); N=53 | -74.1 [-100.0 to 3160.7]

11. Secondary Outcome: Percentage of Participants Who Experienced 50% or More Decrease in Seizure Frequency Over the Perampanel Duration Exposure (Extension Phase)
Description: A responder was a participant who experienced a 50% or greater reduction in seizure frequency per 28 days from pre-perampanel. The percentage of responders from Week 1 of perampanel treatment through successive 13-week intervals (Weeks 1 to 13 for subjects with any data, Weeks 1 to 26 for subjects with exposure of more than 13 weeks, Weeks 1 to 39 for subjects with exposure of more than 26 weeks, and Week 1 to 52 for subjects with exposure of more than 52 weeks) are presented. The perampanel exposure duration starts from the first perampanel dose (in the Core Study for subjects previously randomized to perampanel or Extension Phase for subjects previously randomized to placebo) to the last perampanel dose in the Extension Phase.
Time Frame: Week 1-13, Week 14-26, Week 27-39, and Week 40-52
Population: FAS for Efficacy (Extension Phase)
Measure: Number; unit: Percentage of Participants
Arm/Group | Perampanel (Extension Phase)
Number analyzed (Participants) | 114
Percentage of Participants
  Week 1-13 (any exposure duration); N=114: number analyzed (Participants) | 62
  Week 1-13 (any exposure duration); N=114 | 54.4
  Week 1-13 (at least 13 weeks of exposure); N=109: number analyzed (Participants) | 60
  Week 1-13 (at least 13 weeks of exposure); N=109 | 55.0
  Week 1-13 (at least 26 weeks of exposure); N=107: number analyzed (Participants) | 60
  Week 1-13 (at least 26 weeks of exposure); N=107 | 56.1
  Week 1-13 (at least 39 weeks of exposure); N=90: number analyzed (Participants) | 46
  Week 1-13 (at least 39 weeks of exposure); N=90 | 51.1
  Week 1-13 (at least 52 weeks of exposure); N=67: number analyzed (Participants) | 36
  Week 1-13 (at least 52 weeks of exposure); N=67 | 53.7
  Week 14-26 (at least 26 weeks of exposure); N=107: number analyzed (Participants) | 64
  Week 14-26 (at least 26 weeks of exposure); N=107 | 59.8
  Week 14-26 (at least 39 weeks of exposure); N=90: number analyzed (Participants) | 51
  Week 14-26 (at least 39 weeks of exposure); N=90 | 56.7
  Week 14-26 (at least 52 weeks of exposure); N=67: number analyzed (Participants) | 37
  Week 14-26 (at least 52 weeks of exposure); N=67 | 55.2
  Week 27-39 (at least 39 weeks of exposure); N=90: number analyzed (Participants) | 53
  Week 27-39 (at least 39 weeks of exposure); N=90 | 58.9
  Week 27-39 (at least 52 weeks of exposure); N=67: number analyzed (Participants) | 42
  Week 27-39 (at least 52 weeks of exposure); N=67 | 62.7
  Week 40-52 (at least 52 weeks of exposure); N=53: number analyzed (Participants) | 35
  Week 40-52 (at least 52 weeks of exposure); N=53 | 66.0

12. Secondary Outcome: Mean Change From Baseline to End of Treatment in Cognition Drug Research (CDR) System Global Cognition Score (Extension Phase)
Description: The CDR System Global Cognitive was derived from the average of 5 CDR System cognitive domain scores (Power of Attention, Continuity of Attention, Quality of Episodic Memory, Quality of Working Memory, and Speed of Memory). Domain scores were normalized to mean of 50 and standard deviation of 10 before taking the average. The scale ranged from 0 to 100. An increase in the Global Cognitive Score indicates improvement, while a decrease indicates worsening in cognitive function. The perampanel exposure duration starts from the first perampanel dose (in the Core Study for subjects previously randomized to perampanel or Extension Phase for subjects previously randomized to placebo) to the last perampanel dose in the Extension Phase.
Time Frame: Baseline, Week 9, Week 19, Week, 30, Week 39, Week 52, and End of Treatment (defined as the last nonmissing value after date of first perampanel dose up to 14 days after date of last dose)
Population: The Full Analysis Set for Cognition consisted of all randomized subjects who received study drug in the Extension Phase, had baseline cognition data, and had at least 1 postdose CDR System cognitive test battery assessment after Week 27.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Perampanel (Extension Phase)
Number analyzed (Participants) | 112
Scores on a scale
  Change from Baseline at Week 9 | -3.8 (9.92)
  Change from Baseline at Week 19: number analyzed (Participants) | 105
  Change from Baseline at Week 19 | -1.1 (8.16)
  Change from Baseline at Week 30: number analyzed (Participants) | 105
  Change from Baseline at Week 30 | -1.3 (9.41)
  Change from Baseline at Week 39: number analyzed (Participants) | 73
  Change from Baseline at Week 39 | -2.2 (10.22)
  Change from Baseline at Week 52: number analyzed (Participants) | 63
  Change from Baseline at Week 52 | -0.2 (10.5)
  Change from Baseline at End of Treatment | -1.0 (9.91)

13. Secondary Outcome: Mean Change From Baseline in CDR System Global Cognition Score Over Time (Extension Phase)
Description: The CDR System Global Cognitive was derived from the average of 5 CDR System cognitive domain scores (Power of Attention, Continuity of Attention, Quality of Episodic Memory, Quality of Working Memory, and Speed of Memory). Domain scores were normalized to mean of 50 and SD of 10 before taking the average. The scale ranged from 0 to 100. An increase in the Global Cognitive Score indicates improvement, while a decrease indicates worsening in cognitive function. The data is presented as CDR System Global Cognitive scores at specific intervals (Week 9 for subjects with exposure of more than 9 weeks, Week 19 for subjects with exposure of more than 19 weeks, Week 30 for subjects with exposure of more than 26 weeks, Week 39 for subjects with exposure of more than 39 weeks, and Week 52 for subjects with exposure of more than 52 weeks).
Time Frame: Baseline, Week 9, Week 19, Week, 30, Week 39, and Week 52
Population: FAS for Cognition (Extension Phase)
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Perampanel (Extension Phase)
Number analyzed (Participants) | 112
Scores on a scale
  Week 9 (at least 9 weeks of exposure); N=109: number analyzed (Participants) | 109
  Week 9 (at least 9 weeks of exposure); N=109 | -3.9 (10.03)
  Week 9 (at least 19 weeks of exposure); N=107: number analyzed (Participants) | 107
  Week 9 (at least 19 weeks of exposure); N=107 | -3.7 (9.74)
  Week 9 (at least 26 weeks of exposure); N=107: number analyzed (Participants) | 107
  Week 9 (at least 26 weeks of exposure); N=107 | -3.7 (9.74)
  Week 9 (at least 39 weeks of exposure); N=90: number analyzed (Participants) | 90
  Week 9 (at least 39 weeks of exposure); N=90 | -2.6 (8.73)
  Week 9 (at least 52 weeks of exposure); N=67: number analyzed (Participants) | 67
  Week 9 (at least 52 weeks of exposure); N=67 | -3.1 (8.41)
  Week 19 (at least 19 weeks of exposure); N=105: number analyzed (Participants) | 105
  Week 19 (at least 19 weeks of exposure); N=105 | -1.1 (8.16)
  Week 19 (at least 26 weeks of exposure); N=105: number analyzed (Participants) | 105
  Week 19 (at least 26 weeks of exposure); N=105 | -1.1 (8.16)
  Week 19 (at least 39 weeks of exposure); N=88: number analyzed (Participants) | 88
  Week 19 (at least 39 weeks of exposure); N=88 | -0.8 (8.45)
  Week 19 (at least 52 weeks of exposure); N=65: number analyzed (Participants) | 65
  Week 19 (at least 52 weeks of exposure); N=65 | -1.3 (8.15)
  Week 30 (at least 26 weeks of exposure); N=105: number analyzed (Participants) | 105
  Week 30 (at least 26 weeks of exposure); N=105 | -1.3 (9.41)
  Week 30 (at least 39 weeks of exposure); N=89: number analyzed (Participants) | 89
  Week 30 (at least 39 weeks of exposure); N=89 | -1.0 (9.25)
  Week 30 (at least 52 weeks of exposure); N=66: number analyzed (Participants) | 66
  Week 30 (at least 52 weeks of exposure); N=66 | -1.1 (9.38)
  Week 39 (at least 39 weeks of exposure); N=72: number analyzed (Participants) | 72
  Week 39 (at least 39 weeks of exposure); N=72 | -2.3 (10.28)
  Week 39 (at least 52 weeks of exposure); N=52: number analyzed (Participants) | 52
  Week 39 (at least 52 weeks of exposure); N=52 | -2.3 (10.23)
  Week 52 (at least 52 weeks of exposure); N=49: number analyzed (Participants) | 49
  Week 52 (at least 52 weeks of exposure); N=49 | -0.6 (9.17)

14. Secondary Outcome: Mean Change From Baseline by Visits in CDR System Domain T-Scores (Extension Phase)
Description: The Cognitive measure scores are presented as T-Scores. T-Scores were normalized standard scores with mean of 50 and SD of 10 with an absolute range of 0-100. The T-Scores are based on the norms from healthy age-matched controls from the CDR System database. Cohen's d-effect sizes were used to estimate the clinical relevance of a change in a parameter. A change in a score of 0.2 SD was defined by Cohen as a small effect size, 0.5 SD a medium effect size and 0.8 SD was considered a large effect size. An increase in the T-scores indicates improvement while a decrease in T-scores indicates worsening. Wk = Week and EOT=End of Treatment. The perampanel exposure duration starts from the first perampanel dose (in the Core Study for subjects previously randomized to perampanel or Extension Phase for subjects previously randomized to placebo) to the last perampanel dose in the Extension Phase.
Time Frame: Baseline, Week 9, Week 19, Week 30, Week 39, Week 52, and EOT (defined as the last nonmissing value after date of first dose up to 14 days after date of last dose)
Population: FAS for cognition (Extension Phase)
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Perampanel (Extension Phase)
Number analyzed (Participants) | 112
T-score
  Power of Attention: Week 9 (N=112) | -12.1 (22.24)
  Power of Attention: Week 19 (N=105): number analyzed (Participants) | 105
  Power of Attention: Week 19 (N=105) | -6.5 (19.39)
  Power of Attention: Week 30 (N=105): number analyzed (Participants) | 105
  Power of Attention: Week 30 (N=105) | -8.5 (23.77)
  Power of Attention: Week 39 (N=73): number analyzed (Participants) | 73
  Power of Attention: Week 39 (N=73) | -11.7 (27.04)
  Power of Attention: Week 52 (N=62): number analyzed (Participants) | 62
  Power of Attention: Week 52 (N=62) | -7.5 (26.4)
  Power of Attention: End of treatment (N=112) | -8 (25.75)
  Continuity of Attention: Week 9 (N=112) | -3.1 (8.99)
  Continuity of Attention: Week 19 (N=105): number analyzed (Participants) | 105
  Continuity of Attention: Week 19 (N=105) | -1.7 (8.1)
  Continuity of Attention: Week 30 (N=105): number analyzed (Participants) | 105
  Continuity of Attention: Week 30 (N=105) | -0.9 (8.44)
  Continuity of Attention: Week 39 (N=73): number analyzed (Participants) | 73
  Continuity of Attention: Week 39 (N=73) | -1.7 (8.16)
  Continuity of Attention: Week 52 (N=62): number analyzed (Participants) | 62
  Continuity of Attention: Week 52 (N=62) | -0.9 (8.97)
  Continuity of Attention: End of treatment (N=112) | -0.9 (7.99)
  Quality of episodic secondary Memory:Wk 9 (N=112) | 1.3 (9.27)
  Quality of episodic secondary Memory:Wk 19 (N=105): number analyzed (Participants) | 105
  Quality of episodic secondary Memory:Wk 19 (N=105) | 3.0 (9.76)
  Quality of episodic secondary Memory:Wk 30 (N=104): number analyzed (Participants) | 104
  Quality of episodic secondary Memory:Wk 30 (N=104) | 2.5 (10.15)
  Quality of episodic secondary Memory:Wk 39 (N=73): number analyzed (Participants) | 73
  Quality of episodic secondary Memory:Wk 39 (N=73) | 1.8 (9.78)
  Quality of episodic secondary Memory:Wk 52 (N=63): number analyzed (Participants) | 63
  Quality of episodic secondary Memory:Wk 52 (N=63) | 2.4 (11.33)
  Quality of episodic secondary Memory: EOT (N=112) | 2 (10)
  Quality of working memory (short term):Wk 9(N=112) | -1.8 (14.81)
  Quality of working memory (short term):Wk19(N=105): number analyzed (Participants) | 105
  Quality of working memory (short term):Wk19(N=105) | 1 (12.61)
  Quality of working memory (short term):Wk30(N=105): number analyzed (Participants) | 105
  Quality of working memory (short term):Wk30(N=105) | 1.4 (11.63)
  Quality of working memory (short term):Wk 39(N=73): number analyzed (Participants) | 73
  Quality of working memory (short term):Wk 39(N=73) | -1.2 (13.31)
  Quality of working memory (short term):Wk 52(N=63): number analyzed (Participants) | 63
  Quality of working memory (short term):Wk 52(N=63) | 1.4 (14.85)
  Quality of working memory (short term):EOT (N=112) | 0.5 (12.85)
  Speed of memory: Week 9 (N=111): number analyzed (Participants) | 111
  Speed of memory: Week 9 (N=111) | -3.5 (21.26)
  Speed of memory: Week 19 (N=105): number analyzed (Participants) | 105
  Speed of memory: Week 19 (N=105) | -1.3 (18.23)
  Speed of memory: Week 30 (N=104): number analyzed (Participants) | 104
  Speed of memory: Week 30 (N=104) | -1.4 (20.63)
  Speed of memory: Week 39 (N=73): number analyzed (Participants) | 73
  Speed of memory: Week 39 (N=73) | 1.8 (25.16)
  Speed of memory: Week 52 (N=63): number analyzed (Participants) | 63
  Speed of memory: Week 52 (N=63) | 3.9 (25.34)
  Speed of memory: Week EOT (N=112) | 1 (22.82)

15. Secondary Outcome: Mean Change From Baseline in CDR System Domain T-Score Over Time: Power of Attention (Extension Phase)
Description: The Cognitive measure scores are presented as T-Scores at specific intervals (Week 9 for subjects with exposure of more than 9 weeks, Week 19 for subjects with exposure of more than 19 weeks, Week 30 for subjects with exposure of more than 26 weeks, Week 39 for subjects with exposure of more than 39 weeks, and Week 52 for subjects with exposure of more than 52 weeks). T-Scores were normalized standard scores with mean of 50 and SD of 10 with an absolute range of 0-100. The T-Scores are based on the norms from healthy age-matched controls from the CDR System database. Cohen's d-effect sizes were used to estimate the clinical relevance of a change in a parameter. A change in a score of 0.2 SD was defined by Cohen as a small effect size, 0.5 SD a medium effect size and 0.8 SD was considered a large effect size. An increase in the T-scores indicates improvement while a decrease in T-scores indicates worsening.
Time Frame: Baseline, Week 9, Week 19, Week 30, Week 39, and Week 52
Population: FAS for cognition (Extension Phase)
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Perampanel (Extension Phase)
Number analyzed (Participants) | 112
T-score
  Week 9 (at least 9 weeks of exposure); N=109: number analyzed (Participants) | 109
  Week 9 (at least 9 weeks of exposure); N=109 | -12.3 (22.47)
  Week 9 (at least 19 weeks of exposure); N=107: number analyzed (Participants) | 107
  Week 9 (at least 19 weeks of exposure); N=107 | -11.7 (22.07)
  Week 9 (at least 26 weeks of exposure); N=107: number analyzed (Participants) | 107
  Week 9 (at least 26 weeks of exposure); N=107 | -11.7 (22.07)
  Week 9 (at least 39 weeks of exposure); N=90: number analyzed (Participants) | 90
  Week 9 (at least 39 weeks of exposure); N=90 | -9.5 (17.49)
  Week 9 (at least 52 weeks of exposure); N=67: number analyzed (Participants) | 67
  Week 9 (at least 52 weeks of exposure); N=67 | -9.2 (18.13)
  Week 19 (at least 19 weeks of exposure); N=105: number analyzed (Participants) | 105
  Week 19 (at least 19 weeks of exposure); N=105 | -6.5 (19.39)
  Week 19 (at least 26 weeks of exposure); N=105: number analyzed (Participants) | 105
  Week 19 (at least 26 weeks of exposure); N=105 | -6.5 (19.39)
  Week 19 (at least 39 weeks of exposure); N=88: number analyzed (Participants) | 88
  Week 19 (at least 39 weeks of exposure); N=88 | -4.9 (18.82)
  Week 19 (at least 52 weeks of exposure); N=65: number analyzed (Participants) | 65
  Week 19 (at least 52 weeks of exposure); N=65 | -5.5 (19.37)
  Week 30 (at least 26 weeks of exposure); N=105: number analyzed (Participants) | 105
  Week 30 (at least 26 weeks of exposure); N=105 | -8.5 (23.77)
  Week 30 (at least 39 weeks of exposure); N=89: number analyzed (Participants) | 89
  Week 30 (at least 39 weeks of exposure); N=89 | -7.9 (21.66)
  Week 30 (at least 52 weeks of exposure); N=66: number analyzed (Participants) | 66
  Week 30 (at least 52 weeks of exposure); N=66 | -7.6 (22.39)
  Week 39 (at least 39 weeks of exposure); N=72: number analyzed (Participants) | 72
  Week 39 (at least 39 weeks of exposure); N=72 | -11.8 (27.22)
  Week 39 (at least 52 weeks of exposure); N=52: number analyzed (Participants) | 52
  Week 39 (at least 52 weeks of exposure); N=52 | -12.3 (28.34)
  Week 52 (at least 52 weeks of exposure); N=48: number analyzed (Participants) | 48
  Week 52 (at least 52 weeks of exposure); N=48 | -8.9 (25.45)

16. Secondary Outcome: Mean Change From Baseline in CDR System Domain T-Score Over Time: Continuity of Attention (Extension Phase)
Description: as for outcome 15
Time Frame: Baseline, Week 9, Week 19, Week, 30, Week 39, and Week 52
Population: FAS for cognition (Extension Phase)
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Perampanel (Extension Phase)
Number analyzed (Participants) | 112
T-score
  Week 9 (at least 9 weeks of exposure); N=109: number analyzed (Participants) | 109
  Week 9 (at least 9 weeks of exposure); N=109 | -3.1 (9.11)
  Week 9 (at least 19 weeks of exposure); N=107: number analyzed (Participants) | 107
  Week 9 (at least 19 weeks of exposure); N=107 | -3 (9.01)
  Week 9 (at least 26 weeks of exposure); N=107: number analyzed (Participants) | 107
  Week 9 (at least 26 weeks of exposure); N=107 | -3 (9.01)
  Week 9 (at least 39 weeks of exposure); N=90: number analyzed (Participants) | 90
  Week 9 (at least 39 weeks of exposure); N=90 | -2.8 (9.17)
  Week 9 (at least 52 weeks of exposure); N=67: number analyzed (Participants) | 67
  Week 9 (at least 52 weeks of exposure); N=67 | -3.6 (9.53)
  Week 19 (at least 19 weeks of exposure); N=105: number analyzed (Participants) | 105
  Week 19 (at least 19 weeks of exposure); N=105 | -1.7 (8.1)
  Week 19 (at least 26 weeks of exposure); N=105: number analyzed (Participants) | 105
  Week 19 (at least 26 weeks of exposure); N=105 | -1.7 (8.1)
  Week 19 (at least 39 weeks of exposure); N=88: number analyzed (Participants) | 88
  Week 19 (at least 39 weeks of exposure); N=88 | -1.7 (8.1)
  Week 19 (at least 52 weeks of exposure); N=65: number analyzed (Participants) | 65
  Week 19 (at least 52 weeks of exposure); N=65 | -2.3 (8.49)
  Week 30 (at least 26 weeks of exposure); N=105: number analyzed (Participants) | 105
  Week 30 (at least 26 weeks of exposure); N=105 | -0.9 (8.44)
  Week 30 (at least 39 weeks of exposure); N=89: number analyzed (Participants) | 89
  Week 30 (at least 39 weeks of exposure); N=89 | -1.1 (8.65)
  Week 30 (at least 52 weeks of exposure); N=66: number analyzed (Participants) | 66
  Week 30 (at least 52 weeks of exposure); N=66 | -1.0 (7.47)
  Week 39 (at least 39 weeks of exposure); N=72: number analyzed (Participants) | 72
  Week 39 (at least 39 weeks of exposure); N=72 | -1.8 (8.2)
  Week 39 (at least 52 weeks of exposure); N=52: number analyzed (Participants) | 52
  Week 39 (at least 52 weeks of exposure); N=52 | -1.4 (8.24)
  Week 52 (at least 52 weeks of exposure); N=48: number analyzed (Participants) | 48
  Week 52 (at least 52 weeks of exposure); N=48 | -0.5 (8.6)

17. Secondary Outcome: Mean Change From Baseline in CDR System Domain T-Score Over Time: Quality of Episodic Secondary Memory (Extension Phase)
Description: as for outcome 15
Time Frame: Baseline, Week 9, Week 19, Week 30, Week 39, and Week 52
Population: FAS for cognition (Extension Phase)
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Perampanel (Extension Phase)
Number analyzed (Participants) | 112
T-score
  Week 9 (at least 9 weeks of exposure); N=109: number analyzed (Participants) | 109
  Week 9 (at least 9 weeks of exposure); N=109 | 1.2 (9.35)
  Week 9 (at least 19 weeks of exposure); N=107: number analyzed (Participants) | 107
  Week 9 (at least 19 weeks of exposure); N=107 | 1.4 (9.37)
  Week 9 (at least 26 weeks of exposure); N=107: number analyzed (Participants) | 107
  Week 9 (at least 26 weeks of exposure); N=107 | 1.4 (9.37)
  Week 9 (at least 39 weeks of exposure); N=90: number analyzed (Participants) | 90
  Week 9 (at least 39 weeks of exposure); N=90 | 1.9 (9.67)
  Week 9 (at least 52 weeks of exposure); N=67: number analyzed (Participants) | 67
  Week 9 (at least 52 weeks of exposure); N=67 | 2.0 (10.13)
  Week 19 (at least 19 weeks of exposure); N=105: number analyzed (Participants) | 105
  Week 19 (at least 19 weeks of exposure); N=105 | 3.0 (9.76)
  Week 19 (at least 26 weeks of exposure); N=105: number analyzed (Participants) | 105
  Week 19 (at least 26 weeks of exposure); N=105 | 3.0 (9.76)
  Week 19 (at least 39 weeks of exposure); N=88: number analyzed (Participants) | 88
  Week 19 (at least 39 weeks of exposure); N=88 | 2.8 (9.66)
  Week 19 (at least 52 weeks of exposure); N=65: number analyzed (Participants) | 65
  Week 19 (at least 52 weeks of exposure); N=65 | 2.6 (9.33)
  Week 30 (at least 26 weeks of exposure); N=104: number analyzed (Participants) | 104
  Week 30 (at least 26 weeks of exposure); N=104 | 2.5 (10.15)
  Week 30 (at least 39 weeks of exposure); N=88: number analyzed (Participants) | 88
  Week 30 (at least 39 weeks of exposure); N=88 | 2.5 (10.56)
  Week 30 (at least 52 weeks of exposure); N=65: number analyzed (Participants) | 65
  Week 30 (at least 52 weeks of exposure); N=65 | 2.3 (10.85)
  Week 39 (at least 39 weeks of exposure); N=72: number analyzed (Participants) | 72
  Week 39 (at least 39 weeks of exposure); N=72 | 1.9 (9.85)
  Week 39 (at least 52 weeks of exposure); N=52: number analyzed (Participants) | 52
  Week 39 (at least 52 weeks of exposure); N=52 | 2.9 (10.06)
  Week 52 (at least 52 weeks of exposure); N=49: number analyzed (Participants) | 49
  Week 52 (at least 52 weeks of exposure); N=49 | 2.0 (11.61)

18. Secondary Outcome: Mean Change From Baseline in CDR System Domain T-Score Over Time: Quality of Working Memory (Short Term) (Extension Phase)
Description: The cognitive measure scores are presented as T-Scores at specific intervals (Week 9 for participants with exposure of more than 9 weeks, Week 19 for participants with exposure of more than 19 weeks, Week 30 for participants with exposure of more than 26 weeks, Week 39 for participants with exposure of more than 39 weeks, and Week 52 for participants with exposure of more than 52 weeks). T-Scores were normalized standard scores with mean of 50 and SD of 10 with an absolute range of 0-100. The T-Scores are based on the norms from healthy age-matched controls from the CDR System database. Cohen's d-effect sizes were used to estimate the clinical relevance of a change in a parameter. A change in a score of 0.2 SD was defined by Cohen as a small effect size, 0.5 SD a medium effect size and 0.8 SD was considered a large effect size. An increase in the T-scores indicates improvement while a decrease in T-scores indicates worsening.
Time Frame: Baseline, Week 9, Week 19, Week, 30, Week 39, and Week 52
Population: FAS for cognition (Extension Phase)
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Perampanel (Extension Phase)
Number analyzed (Participants) | 112
T-score
  Week 9 (at least 9 weeks of exposure); N=109: number analyzed (Participants) | 109
  Week 9 (at least 9 weeks of exposure); N=109 | -2.0 (14.95)
  Week 9 (at least 19 weeks of exposure); N=107: number analyzed (Participants) | 107
  Week 9 (at least 19 weeks of exposure); N=107 | -1.9 (14.93)
  Week 9 (at least 26 weeks of exposure); N=107: number analyzed (Participants) | 107
  Week 9 (at least 26 weeks of exposure); N=107 | -1.9 (14.93)
  Week 9 (at least 39 weeks of exposure); N=90: number analyzed (Participants) | 90
  Week 9 (at least 39 weeks of exposure); N=90 | -1.2 (14.58)
  Week 9 (at least 52 weeks of exposure); N=67: number analyzed (Participants) | 67
  Week 9 (at least 52 weeks of exposure); N=67 | -0.6 (12.03)
  Week 19 (at least 19 weeks of exposure); N=105: number analyzed (Participants) | 105
  Week 19 (at least 19 weeks of exposure); N=105 | 1.0 (12.61)
  Week 19 (at least 26 weeks of exposure); N=105: number analyzed (Participants) | 105
  Week 19 (at least 26 weeks of exposure); N=105 | 1.0 (12.61)
  Week 19 (at least 39 weeks of exposure); N=88: number analyzed (Participants) | 88
  Week 19 (at least 39 weeks of exposure); N=88 | 1.0 (12.24)
  Week 19 (at least 52 weeks of exposure); N=65: number analyzed (Participants) | 65
  Week 19 (at least 52 weeks of exposure); N=65 | 1.1 (8.91)
  Week 30 (at least 26 weeks of exposure); N=105: number analyzed (Participants) | 105
  Week 30 (at least 26 weeks of exposure); N=105 | 1.4 (11.63)
  Week 30 (at least 39 weeks of exposure); N=89: number analyzed (Participants) | 89
  Week 30 (at least 39 weeks of exposure); N=89 | 1.5 (11.64)
  Week 30 (at least 52 weeks of exposure); N=66: number analyzed (Participants) | 66
  Week 30 (at least 52 weeks of exposure); N=66 | 1.1 (10.00)
  Week 39 (at least 39 weeks of exposure); N=72: number analyzed (Participants) | 72
  Week 39 (at least 39 weeks of exposure); N=72 | -1.1 (13.38)
  Week 39 (at least 52 weeks of exposure); N=52: number analyzed (Participants) | 52
  Week 39 (at least 52 weeks of exposure); N=52 | -0.1 (11.77)
  Week 52 (at least 52 weeks of exposure); N=49: number analyzed (Participants) | 49
  Week 52 (at least 52 weeks of exposure); N=49 | 2.9 (10.22)

19. Secondary Outcome: Mean Change From Baseline in CDR System Domain T-Score Over Time: Speed of Memory (Extension Phase)
Description: as for outcome 15
Time Frame: Baseline, Week 9, Week 19, Week, 30, Week 39, and Week 52
Population: FAS for cognition (Extension Phase)
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Perampanel (Extension Phase)
Number analyzed (Participants) | 112
T-score
  Week 9 (at least 9 weeks of exposure); N=108: number analyzed (Participants) | 108
  Week 9 (at least 9 weeks of exposure); N=108 | -3.7 (21.51)
  Week 9 (at least 19 weeks of exposure); N=106: number analyzed (Participants) | 106
  Week 9 (at least 19 weeks of exposure); N=106 | -3.1 (21.31)
  Week 9 (at least 26 weeks of exposure); N=106: number analyzed (Participants) | 106
  Week 9 (at least 26 weeks of exposure); N=106 | -3.1 (21.31)
  Week 9 (at least 39 weeks of exposure); N=89: number analyzed (Participants) | 89
  Week 9 (at least 39 weeks of exposure); N=89 | -1.6 (20.85)
  Week 9 (at least 52 weeks of exposure); N=67: number analyzed (Participants) | 67
  Week 9 (at least 52 weeks of exposure); N=67 | -4.3 (15.34)
  Week 19 (at least 19 weeks of exposure); N=105: number analyzed (Participants) | 105
  Week 19 (at least 19 weeks of exposure); N=105 | -1.3 (18.23)
  Week 19 (at least 26 weeks of exposure); N=105: number analyzed (Participants) | 105
  Week 19 (at least 26 weeks of exposure); N=105 | -1.3 (18.23)
  Week 19 (at least 39 weeks of exposure); N=88: number analyzed (Participants) | 88
  Week 19 (at least 39 weeks of exposure); N=88 | -1.1 (18.31)
  Week 19 (at least 52 weeks of exposure); N=65: number analyzed (Participants) | 65
  Week 19 (at least 52 weeks of exposure); N=65 | -2.4 (15.57)
  Week 30 (at least 26 weeks of exposure); N=104: number analyzed (Participants) | 104
  Week 30 (at least 26 weeks of exposure); N=104 | -1.4 (20.63)
  Week 30 (at least 39 weeks of exposure); N=88: number analyzed (Participants) | 88
  Week 30 (at least 39 weeks of exposure); N=88 | -0.7 (19.74)
  Week 30 (at least 52 weeks of exposure); N=65: number analyzed (Participants) | 65
  Week 30 (at least 52 weeks of exposure); N=65 | -1.0 (20.06)
  Week 39 (at least 39 weeks of exposure); N=72: number analyzed (Participants) | 72
  Week 39 (at least 39 weeks of exposure); N=72 | 1.6 (25.29)
  Week 39 (at least 52 weeks of exposure); N=52: number analyzed (Participants) | 52
  Week 39 (at least 52 weeks of exposure); N=52 | -0.5 (24.97)
  Week 52 (at least 52 weeks of exposure); N=49: number analyzed (Participants) | 49
  Week 52 (at least 52 weeks of exposure); N=49 | 1.8 (24.05)

20. Secondary Outcome: Change From Baseline to End of Treatment in Controlled Oral Word Association Test Scores (COWAT) (Extension Phase)
Description: The COWAT test measured the executive function of the frontal lobe and consisted of examinations of category/meaning fluency and letter/phoneme fluency. It consisted of 2 parts which included the Letter Fluency task and the Category Fluency task. For the Letter Fluency task, the participant was given one minute to list as many words as they could which began with a given letter from the following set of 3 letters: F, A, and L. The number of correct words from the 3 sets comprised the Letter Fluency score. For the Category Fluency task, the participant was given one minute to list as many words as they could which belonged to a given category. The number of correct words comprised the Category Fluency score. Total score was calculated as sum of acceptable words generated. The scale ranged from 0-90, with higher scores indicating improvement in language.
Time Frame: From Baseline up to Week 52 or up to EOT (defined as the last nonmissing value after date of first dose up to 14 days after date of last dose)
Population: FAS for cognition (Extension Phase)
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Perampanel (Extension Phase)
Number analyzed (Participants) | 112
Scores on a scale
  Letter Fluency Score; N=110: number analyzed (Participants) | 110
  Letter Fluency Score; N=110 | 2.2 (7.98)
  Category Fluency Score; N=110: number analyzed (Participants) | 110
  Category Fluency Score; N=110 | -0.3 (4.02)

21. Secondary Outcome: Change From Baseline to End of Treatment in Time to Complete Lafayette Grooved Pegboard Test (LGPT) (Extension Phase)
Description: The LGPT test measured visuomotor skills. This test was a manipulative dexterity test that consisted of a metal matrix of 25 holes with randomly positioned slots. The participant was required to insert 25 grooved pegs into the holes. The task was completed once for each hand; firstly, using the dominant hand followed by the non-dominant hand. The task was timed and the scores were the time taken for the participant to complete all 25 pegs for each hand. If the test cannot be completed within 300 seconds, 300 seconds were recorded for the time. An increase in score (longer time) indicated worsening of visuomotor skills. The time to complete test is presented as mean seconds +/- SD.
Time Frame: as for outcome 20
Population: FAS for cognition (Extension Phase)
Measure: Mean (Standard Deviation); unit: Seconds
Arm/Group | Perampanel (Extension Phase)
Number analyzed (Participants) | 112
Seconds
  Dominant Hand | 0.5 (18.67)
  Non-Dominant Hand | -3.3 (22.49)

22. Secondary Outcome: Mean Change From Baseline in Bone Age Minus Age (Months) From Hand X-ray (Extension Phase)
Description: Bone age was measured using hand X-ray. The mean change from Baseline in bone age (months) minus age (months) from the hand x-ray was assessed. "+" means bone age is older than age and "-" means bone age is younger than age.
Time Frame: as for outcome 20
Population: The Safety Analysis Set consisted of all enrolled subjects who (1) took at least 1 dose of perampanel in the Extension Phase and (2) had a safety assessment after the first dose of perampanel in the Extension Phase.
Measure: Mean (Standard Deviation); unit: Months
Arm/Group | Perampanel (Extension Phase)
Number analyzed (Participants) | 114
Months
  Baseline: number analyzed (Participants) | 110
  Baseline | 3.3 (16.21)
  Change from Baseline at EOT: number analyzed (Participants) | 109
  Change from Baseline at EOT | -2.0 (9.83)

23. Secondary Outcome: Change From Baseline to End of Treatment (EOT) for the Tanner Stage
Description: The effect of perampanel on growth and development in adolescents (male and female), including sexual development was measured using Tanner scale. The scale defined physical measurements of development based on external primary and secondary sex characteristics, such as the size of the breasts, genitals, testicular volume and development of pubic hair. Tanner scale consisted of 5 scales from I to V (1: pre-pubertal to 5: adult). Data is reported as the change from Baseline to End of Treatment for the Tanner Stage.
Time Frame: From Baseline up to Week 52 or EOT (defined as the last nonmissing value after date of first dose up to 14 days after date of last dose)
Population: SAS (Extension Phase)
Measure: Number; unit: participants
Arm/Group | Perampanel (Extension Phase)
Number analyzed (Participants) | 112
participants
  Baseline Tanner stage II to EOT Tanner stage II | 5
  Baseline Tanner stage II to EOT Tanner stage III | 2
  Baseline Tanner stage II to EOT Tanner stage IV | 3
  Baseline Tanner stage III to EOT Tanner stage III | 8
  Baseline Tanner stage III to EOT Tanner stage IV | 12
  Baseline Tanner stage III to EOT Tanner stage V | 3
  Baseline Tanner stage IV to EOT Tanner stage IV | 22
  Baseline Tanner stage IV to EOT Tanner stage V | 19
  Baseline Tanner stage V to EOT Tanner stage V | 40

ADVERSE EVENTS:
Time Frame: From start of first dose of study drug up to approximately 23 weeks for the Core Study and up to approximately 83 weeks for the extension phase.
Description: Data are presented as treatment emergent adverse events (TEAEs), defined as an adverse event that started/increased in severity on/after the first dose of study medication up to 30 days after the final dose of study medication. Safety Analysis Set (SAS), defined as all subjects who took ≥ 1 study drug dose and had a postbaseline safety assessment.
Arm/Group | Perampanel (Core Study) | Placebo (Core Study) | Perampanel (Extension Phase)
Serious Adverse Events (participants affected / at risk) | 5/85 | 2/48 | 19/114
Other Adverse Events (participants affected / at risk) | 67/85 | 30/48 | 95/114
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Perampanel (Core Study) (N=85) | Placebo (Core Study) (N=48) | Perampanel (Extension Phase) (N=114)
Foot fracture (Injury, poisoning and procedural complications) | 1 | 0 | 1
Accidental overdose (Injury, poisoning and procedural complications) | 0 | 0 | 1
Intentional overdose (Injury, poisoning and procedural complications) | 0 | 0 | 1
Hand fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Ligament rupture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Influenza (Infections and infestations) | 0 | 1 | 0
Nasopharyngitis (Infections and infestations) | 1 | 0 | 1
Convulsion (Nervous system disorders) | 0 | 1 | 4
Partial seizures with secondary generalisation (Nervous system disorders) | 1 | 0 | 1
Simple partial seizures (Nervous system disorders) | 0 | 0 | 1
Status epilepticus (Nervous system disorders) | 0 | 0 | 1
Aggression (Psychiatric disorders) | 2 | 0 | 4
Suicidal ideation (Psychiatric disorders) | 0 | 0 | 1
Suicide attempt (Psychiatric disorders) | 0 | 0 | 1
Gastroduodenitis (Gastrointestinal disorders) | 1 | 0 | 1
Testicular necrosis (Reproductive system and breast disorders) | 0 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Perampanel (Core Study) (N=85) | Placebo (Core Study) (N=48) | Perampanel (Extension Phase) (N=114)
Pituitary tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Multiple allergies (Immune system disorders) | 1 | 0 | 1
Drug hypersensitivity (Immune system disorders) | 0 | 0 | 1
Asthenia (General disorders) | 0 | 2 | 2
Fatigue (General disorders) | 8 | 1 | 13
Local swelling (General disorders) | 1 | 0 | 1
Pyrexia (General disorders) | 2 | 1 | 8
Gait disturbance (General disorders) | 0 | 0 | 1
Irritability (General disorders) | 6 | 1 | 7
Adjustment disorder (Psychiatric disorders) | 1 | 0 | 0
Aggression (Psychiatric disorders) | 6 | 1 | 10
Anger (Psychiatric disorders) | 2 | 0 | 2
Anxiety (Psychiatric disorders) | 1 | 0 | 1
Bradyphrenia (Psychiatric disorders) | 3 | 0 | 3
Confusional state (Psychiatric disorders) | 3 | 0 | 3
Depressed mood (Psychiatric disorders) | 1 | 0 | 1
Euphoric mood (Psychiatric disorders) | 2 | 1 | 2
Initial insomnia (Psychiatric disorders) | 0 | 1 | 1
Insomnia (Psychiatric disorders) | 3 | 3 | 5
Intentional self-injury (Psychiatric disorders) | 1 | 0 | 0
Mood altered (Psychiatric disorders) | 2 | 1 | 1
Mood swings (Psychiatric disorders) | 3 | 1 | 4
Self-injurious ideation (Psychiatric disorders) | 1 | 0 | 1
Tearfulness (Psychiatric disorders) | 0 | 1 | 0
Abnormal Behaviour (Psychiatric disorders) | 0 | 0 | 1
Daydreaming (Psychiatric disorders) | 0 | 0 | 1
Depression (Psychiatric disorders) | 0 | 0 | 1
Nervousness (Psychiatric disorders) | 0 | 0 | 3
Regressive behaviour (Psychiatric disorders) | 0 | 0 | 1
Somnambulism (Psychiatric disorders) | 0 | 0 | 1
Menstruation irregular (Reproductive system and breast disorders) | 1 | 0 | 1
Testicular torsion (Reproductive system and breast disorders) | 0 | 0 | 1
Concussion (Injury, poisoning and procedural complications) | 1 | 0 | 2
Contusion (Injury, poisoning and procedural complications) | 3 | 0 | 3
Excoriation (Injury, poisoning and procedural complications) | 2 | 0 | 2
Joint injury (Injury, poisoning and procedural complications) | 1 | 0 | 0
Laceration (Injury, poisoning and procedural complications) | 1 | 0 | 1
Ligament rupture (Injury, poisoning and procedural complications) | 1 | 0 | 1
Muscle strain (Injury, poisoning and procedural complications) | 1 | 0 | 1
Radius fracture (Injury, poisoning and procedural complications) | 0 | 1 | 1
Tongue injury (Injury, poisoning and procedural complications) | 0 | 1 | 0
Wrist fracture (Injury, poisoning and procedural complications) | 1 | 0 | 1
Accidental Overdose (Injury, poisoning and procedural complications) | 0 | 0 | 2
Animal Bite (Injury, poisoning and procedural complications) | 0 | 0 | 2
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 1
Foot fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Hand fracture (Injury, poisoning and procedural complications) | 0 | 0 | 2
Head Injury (Injury, poisoning and procedural complications) | 0 | 0 | 2
Limb Injury (Injury, poisoning and procedural complications) | 0 | 0 | 1
Sunburn (Injury, poisoning and procedural complications) | 0 | 0 | 1
Blood creatine phosphokinase increased (Investigations) | 3 | 2 | 4
Blood pressure diastolic decreased (Investigations) | 0 | 1 | 0
Platelet count decreased (Investigations) | 1 | 0 | 0
Thyroxine decreased (Investigations) | 0 | 1 | 1
Weight decreased (Investigations) | 0 | 1 | 1
Weight increased (Investigations) | 5 | 0 | 8
White blood cell count decreased (Investigations) | 1 | 0 | 1
Alanine aminotransferase increased (Investigations) | 0 | 0 | 2
Aspartate Aminotransferase Increased (Investigations) | 0 | 0 | 2
Blood Cholesterol Increased (Investigations) | 0 | 0 | 1
Blood Glucose Decreased (Investigations) | 0 | 0 | 1
Blood Pressure Decreased (Investigations) | 0 | 0 | 1
Blood Sodium Increased (Investigations) | 0 | 0 | 1
Blood Triglycerides Increased (Investigations) | 0 | 0 | 1
Electrocardiogram T Wave Abnormal (Investigations) | 0 | 0 | 1
Bradycardia (Cardiac disorders) | 1 | 0 | 3
Angina pectoris (Cardiac disorders) | 0 | 0 | 1
Sinus bradycardia (Cardiac disorders) | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 2
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 2
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Diaphragmatic Spasm (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Snoring (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Eosinophilia (Blood and lymphatic system disorders) | 1 | 2 | 3
Monocytosis (Blood and lymphatic system disorders) | 0 | 1 | 1
Neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 0
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 2
Leukopenia (Blood and lymphatic system disorders) | 1 | 0 | 1
Ataxia (Nervous system disorders) | 4 | 0 | 5
Balance disorder (Nervous system disorders) | 2 | 0 | 3
Clumsiness (Nervous system disorders) | 2 | 0 | 2
Cognitive disorder (Nervous system disorders) | 0 | 1 | 2
Convulsion (Nervous system disorders) | 4 | 4 | 10
Depressed level of consciousness (Nervous system disorders) | 1 | 0 | 0
Disturbance in attention (Nervous system disorders) | 2 | 0 | 2
Dizziness (Nervous system disorders) | 26 | 7 | 34
Drooling (Nervous system disorders) | 1 | 0 | 1
Dysarthria (Nervous system disorders) | 1 | 0 | 2
Headache (Nervous system disorders) | 9 | 7 | 13
Hypoaesthesia (Nervous system disorders) | 1 | 0 | 1
Hypotonia (Nervous system disorders) | 1 | 0 | 1
Lethargy (Nervous system disorders) | 2 | 0 | 4
Memory impairment (Nervous system disorders) | 1 | 0 | 1
Partial seizures with secondary generalisation (Nervous system disorders) | 0 | 1 | 0
Simple partial seizures (Nervous system disorders) | 1 | 1 | 3
Slow speech (Nervous system disorders) | 2 | 0 | 2
Somnolence (Nervous system disorders) | 13 | 2 | 22
Syncope (Nervous system disorders) | 1 | 0 | 2
Tremor (Nervous system disorders) | 1 | 0 | 3
Aphasia (Nervous system disorders) | 0 | 0 | 2
Complex Partial Seizures (Nervous system disorders) | 0 | 0 | 1
Coordination Abnormal (Nervous system disorders) | 0 | 0 | 1
Dyskinesia (Nervous system disorders) | 0 | 0 | 1
Dyspraxia (Nervous system disorders) | 0 | 0 | 1
Epilepsy (Nervous system disorders) | 0 | 0 | 3
Migraine (Nervous system disorders) | 0 | 0 | 1
Partial Seizures (Nervous system disorders) | 0 | 0 | 1
Postictal Headache (Nervous system disorders) | 0 | 0 | 1
Diplopia (Eye disorders) | 0 | 1 | 2
Mydriasis (Eye disorders) | 1 | 0 | 1
Vision blurred (Eye disorders) | 3 | 0 | 2
Visual impairment (Eye disorders) | 1 | 0 | 1
Myopia (Eye disorders) | 0 | 0 | 1
Visual acuity reduced (Eye disorders) | 0 | 0 | 1
Vertigo (Ear and labyrinth disorders) | 0 | 1 | 6
Tinnitus (Ear and labyrinth disorders) | 1 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 2 | 2
Abdominal pain upper (Gastrointestinal disorders) | 4 | 1 | 4
Constipation (Gastrointestinal disorders) | 1 | 1 | 1
Diarrhoea (Gastrointestinal disorders) | 2 | 1 | 4
Gastritis (Gastrointestinal disorders) | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 2 | 2 | 6
Abdominal discomfort (Gastrointestinal disorders) | 2 | 0 | 2
Dry mouth (Gastrointestinal disorders) | 1 | 0 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0 | 1
Hyperchlorhydria (Gastrointestinal disorders) | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 2 | 0 | 2
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 1
Enterocolitis (Gastrointestinal disorders) | 0 | 0 | 1
Toothache (Gastrointestinal disorders) | 0 | 0 | 1
Haematuria (Renal and urinary disorders) | 1 | 0 | 1
Crystalluria (Renal and urinary disorders) | 0 | 0 | 1
Enuresis (Renal and urinary disorders) | 0 | 0 | 2
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 1 | 1
Dermal cyst (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 | 0 | 2
Heat rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 3
Swelling face (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Acne (Skin and subcutaneous tissue disorders) | 0 | 0 | 2
Dermatitis Acneiform (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Macule (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Rash Maculo-Papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Seborrhoeic Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Epiphyses premature fusion (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Myositis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Appetite disorder (Metabolism and nutrition disorders) | 0 | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 3 | 1 | 4
Hypernatraemia (Metabolism and nutrition disorders) | 1 | 0 | 1
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 1 | 0 | 1
Increased appetite (Metabolism and nutrition disorders) | 4 | 0 | 4
Obesity (Metabolism and nutrition disorders) | 1 | 0 | 1
Bronchitis (Infections and infestations) | 0 | 1 | 3
Fungal skin infection (Infections and infestations) | 1 | 0 | 1
Influenza (Infections and infestations) | 1 | 0 | 2
Nasopharyngitis (Infections and infestations) | 3 | 3 | 13
Pharyngitis (Infections and infestations) | 1 | 0 | 1
Respiratory tract infection (Infections and infestations) | 1 | 0 | 1
Sinusitis (Infections and infestations) | 1 | 1 | 1
Skin infection (Infections and infestations) | 1 | 0 | 1
Tonsillitis (Infections and infestations) | 2 | 0 | 2
Tracheitis (Infections and infestations) | 0 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 4 | 3 | 5
Urinary tract infection (Infections and infestations) | 2 | 1 | 3
Vaginitis bacterial (Infections and infestations) | 1 | 0 | 0
Varicella (Infections and infestations) | 0 | 1 | 0
Viral upper respiratory tract infection (Infections and infestations) | 2 | 0 | 3
Acarodermatitis (Infections and infestations) | 0 | 0 | 1
Cellulitis (Infections and infestations) | 0 | 0 | 1
Cystitis (Infections and infestations) | 0 | 0 | 1
Fungal infection (Infections and infestations) | 0 | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 0 | 2
Laryngitis (Infections and infestations) | 0 | 0 | 1
Localised infection (Infections and infestations) | 0 | 0 | 1
Oral Herpes (Infections and infestations) | 0 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 0 | 1
Rhinitis (Infections and infestations) | 0 | 0 | 1
Viral infection (Infections and infestations) | 0 | 0 | 1
Bacterial vaginosis (Infections and infestations) | 0 | 0 | 1
Miliaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other